CLINICAL TRIAL: NCT02094131
Title: Effects of Training Using Volume and Flow-oriented Incentive Spirometry in Healthy Subjects - Case-control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ivanize Mariana Masselli dos Reis, Specialist, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IMMR-01
Record Dates: First submitted 2014-03-13; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: incentive spirometry; flow-oriented spirometer; volume-oriented spirometer; physical therapy; respiratory muscle training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cliniflo group (CG) (Experimental): Training using flow-oriented incentive spirometry Cliniflo
  Interventions: Other: Cliniflo group (CG)
- Voldyne group (VG) (Experimental): Training using volume-oriented incentive spirometry Voldyne
  Interventions: Other: Voldyne group (VG)
- Control group (CONG) (No Intervention): No intervention. Assessment and reassessment after 5 weeks.

INTERVENTIONS:
Other: Voldyne group (VG) — VG: slow deep breaths through the mouthpiece of the incentive Voldyne5000® were conducted from the tidal volume (TV) until the total lung capacity (TLC), holding the maximum inspiration. All individuals should maintain "yellow cup" ("yellow flow cup") at a range of flow "Best" in as long as possible. The training lasted approximately 50 minutes, were held twice a week on alternate days, for five consecutive weeks, totaling 10 sessions. Performed three sets of 15 repetitions.
  Arms: Voldyne group (VG)
Other: Cliniflo group (CG) — CG: slow deep breaths through the mouthpiece of the incentive Cliniflo® from tidal volume (TV) were performed until the total lung capacity (TLC), holding the maximum inspiration. The volume flow of 100 ml / s for Cliniflo® was standardized, being envisaged to keep the yellow indicator behind the "happy face" for all individuals.The training lasted approximately 50 minutes, were held twice a week on alternate days, for five consecutive weeks, totaling 10 sessions. Performed three sets of 15 repetitions.
  Arms: Cliniflo group (CG)

SUMMARY:
Experimental Procedure: The subjects underwent an initial interview in which was filled in a form of anamnesis, in addition to being assessed and reassessed by spirometry, dynamic circumference and manometer. Moreover, responded international physical activity questionnaire (IPAQ - short version) in order to characterize the physical activity level of each participant being classified as inactive, irregularly active, active, and very active. The same examiner performed the assessments and reassessments of individuals after a training program.

DETAILED DESCRIPTION:
Spirometry: It was performed by a portable spirometer Easy One® , according to the guidelines of the American Thoracic Society / European Respiratory Society (ATS / ERS). The values obtained were compared with the values predicted by Knudson et al..

Cirtometry Dynamics: provided information on the degree of thoracoabdominal mobility and was performed with the use of a tape measure , which was used to measure the chest circumference during maximal inspiratory and expiratory phase . Measurements were taken horizontally at three different levels: axillary, xiphoid and abdominal, taking as references the axillary fold bottom edge of the xiphoid and umbilicus, respectively. Three measurements on each level were performed.

The maximum values of inspiration and expiration were obtained, being considered for analysis, the highest value of the three measurements and subsequently the Index of Amplitude (IA) proposed by Jamami et al. was calculated in order to mitigate the different dimensions of the chest and abdomen.

Respiratory muscle strength : They were taken with the subject in a sitting position using a digital manometer (MVD300 - Globalmed®) calibrated, nose clip, with the nozzle held firmly between his lips.

The maximal inspiratory pressure (MIP) was obtained by a maximal inspiration preceded by a maximal expiration next to the residual volume (RV) , and to measure maximal expiratory pressure (MEP) a maximal inspiration was next performed to capacity total lung (CPT) followed by a maximal expiration.

The evaluation was considered complete when the individual performed three acceptable measures and, among these, a minimum of two reproducible . The last value found could not be superior to the others. Maneuvers with the support pressure by three seconds, and reproducible measurements with a variation less than or equal to 10% of the highest value were considered acceptable. For analysis was considered the greatest pressure value achieved. MIP and MEP obtained the values predicted by the equations of Neder et al. were compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* Spirometric values within normal limits
* Body mass index (BMI) between 18 and 29.9 (kg/m2)
* Without previous or current history of smoking
* Did not report the presence of neuromuscular, respiratory or cardiac disease

Exclusion Criteria:

* Inability to understand and / or perform procedures
* Physically active and very active individuals

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing (Spirometry) | up to 5 weeks
  vital capacity (VC) (%predicted) peak expiratory flow (PEF) (%predicted) forced vital capacity (FVC) (%predicted) forced expiratory volume in one second (FEV1) (%predicted) forced expiratory volume in one second/forced vital capacity ratio (FEV1/FVC) maximum voluntary ventilation (MVV) (%predicted)

SECONDARY OUTCOMES:
Respiratory muscle strength (Maximal inspiratory and expiratory pressures-manometer) | Baseline and 5 weeks
  maximal inspiratory pressure (MIP) (cmH2O) maximal expiratory pressure (MEP) (cmH2O)

OTHER OUTCOMES:
Thoracoabdominal Mobility (Cirtometry Dynamics) | Baseline and 5 weeks
  Amplitude Index axillary (AIA) Amplitude Index xiphoid (AIX) Amplitude Index abdominal (AIAB)

CONTACTS AND LOCATIONS:
Overall Officials: Ivanize Mariana M dos Reis, Specialist, Principal Investigator — Universidade Federal de Sao Carlos; Mauricio Jamami, PhD, Study Director — Universidade Federal de Sao Carlos; Bruna V Pessoa, PhD, Study Chair — Universidade Federal de Sao Carlos
Locations (1):
- Ivanize Mariana Masselli dos Reis, São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Knudson RJ, Lebowitz MD, Holberg CJ, Burrows B. Changes in the normal maximal expiratory flow-volume curve with growth and aging. Am Rev Respir Dis. 1983 Jun;127(6):725-34. doi: 10.1164/arrd.1983.127.6.725. PMID 6859656
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten C, Gustafsson P, Jensen R, Macintyre N, McKay RT, Pedersen OF, Pellegrino R, Viegi G, Wanger J. Standardisation of lung function testing: the authors' replies to readers' comments. Eur Respir J. 2010 Dec;36(6):1496-8. doi: 10.1183/09031936.00130010. No abstract available. PMID 21119213
- [Result] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Result] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Result] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401